CLINICAL TRIAL: NCT00013572
Title: A Phase I Study of Aventis Pasteur Live Recombinant ALVAC-HIV (vCP205, HIV-1 Env/Gag/Pol) in Seronegative Adults Administered (1) Subcutaneously Via Ex Vivo Transfected, Autologous Dendritic Cells, (2) Intradermally, or (3) Intramuscularly
Brief Title: HIV Candidate Vaccine, ALVAC-HIV-1, Administration in HIV-Negative Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Prevention
Other Study IDs: B011; RV 138
Record Dates: First submitted 2001-03-21; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-03

CONDITIONS: HIV Infections; HIV Seronegativity
Keywords: Injections, Intramuscular; Injections, Intradermal; Injections, Subcutaneous; HIV-1; AIDS Vaccines; Dendritic Cells; HIV Seronegativity; Genes, env; Genes, pol; Genes, gag; Transfection; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: ALVAC-HIV MN120TMG (vCP205)

SUMMARY:
The purpose of this study is to determine the best way to administer the candidate HIV vaccine, ALVAC HIV-1 (vCP205).

DETAILED DESCRIPTION:
Healthy adult volunteers are assigned randomly to either a vaccine or placebo group. Injections are received either intramuscularly, intradermally, or by delivery under the skin of the volunteer's own white blood cells which have had dendritic cell reinfusion. Volunteers are vaccinated at 0, 1, 3, and 6 month time points. Volunteers are closely monitored for 1 hour after vaccination and keep a diary of symptoms for 1 week post-immunization. Volunteers undergo leukopheresis at the start of the study and after the last vaccination at Walter Reed Army Medical Center. Volunteers receive compensation benefits.

ELIGIBILITY:
Inclusion Criteria

Volunteers may be eligible for this study if they:

* Are legal US residents.
* Are healthy adults from 18 to 55 years of age.

Exclusion Criteria

Volunteers will not be eligible for this study if they:

* Are HIV-positive.
* Are at highest risk for HIV infection.
* Are pregnant or breast-feeding.
* Are allergic to eggs or neomycin.
* Use certain prescription medications.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36

CONTACTS AND LOCATIONS:
Overall Officials: Mary Marovich, Principal Investigator
Locations (1):
- Walter Reed Army Institute of Research (WRAIR), Rockville, Maryland, United States

REFERENCES:
- [Derived] Eller MA, Slike BM, Cox JH, Lesho E, Wang Z, Currier JR, Darden JM, Polonis VR, Vahey MT, Peel S, Robb ML, Michael NL, Marovich MA. A double-blind randomized phase I clinical trial targeting ALVAC-HIV vaccine to human dendritic cells. PLoS One. 2011;6(9):e24254. doi: 10.1371/journal.pone.0024254. Epub 2011 Sep 16. PMID 21949699